CLINICAL TRIAL: NCT06442566
Title: Sequential Trial of Adding Buprenorphine, Cognitive Behavioral Treatment, and Transcranial Magnetic Stimulation to Improve Outcomes of Long-Term Opioid Therapy for Chronic Pain (ACTION)
Brief Title: ACTION: Trial of Adding Buprenorphine, CBT, and TMS to Improve Outcomes of Long-Term Opioid Therapy for Chronic Pain
Acronym: ACTION
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kelly Barth, Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00130123; 1R01DA058620 (NIH)
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Opioid Withdrawal; Chronic Pain
Keywords: opioids, long-term opioid use, chronic pain, TMS
MeSH Terms: conditions — Chronic Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: SMART
Who Masked: Participant, Investigator
Masking Description: Arm 1 open label, double blind procedures for randomization of BUP and TMS
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- open label BUP (Experimental)
  Interventions: Drug: Buprenorphine Patch
- Real vs Placebo BUP (Active Comparator)
  Interventions: Drug: Buprenorphine Patch; Drug: Placebo
- Real vs Sham TMS (Active Comparator)
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Device: Sham Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Drug: Buprenorphine Patch — Buprenorphine patch dosing will be individualized based on each participant's current morphine-equivalent dose (per package insert/recommendations; between 5mcg and 20mcg per hour). Dosage based on baseline MEQ (<30 MEQ = 5mcg/hr patch, 30-80 MEQ =10-15mcg/hour patch; >80 MEQ = 20mcg/hour patch), which will remain on for 7 days (Phase Ia Days 1-7), as tolerated
  Arms: Real vs Placebo BUP; open label BUP
Drug: Placebo — double-blinded randomization to placebo or transdermal buprenorphine
  Arms: Real vs Placebo BUP
Device: Transcranial Magnetic Stimulation (TMS) — double-blinded randomization to REAL intermittent theta burst (iTBS) rTMS
  Arms: Real vs Sham TMS
Device: Sham Transcranial Magnetic Stimulation (TMS) — double-blinded randomization to SHAM intermittent theta burst (iTBS) rTMS
  Arms: Real vs Sham TMS

SUMMARY:
This study will sequentially evaluate three novel and scalable interventions for at-risk individuals on long term opioid therapy for chronic pain: (1) low-dose transdermal buprenorphine initiation without a period of opioid withdrawal; (2) a brief Cognitive Behavioral Intervention for pain (CBI); and (3) "accelerated" rTMS over the left dorsolateral prefrontal cortex, by examining standardized repeated measures of clinical outcomes at baseline, during treatment, and at 4-, 12-, 24- and 52-week follow-up.

DETAILED DESCRIPTION:
With little evidence available to guide the provision of clinical care for patients on long-term opioid therapy (LTOT) in whom the risks outweigh the benefits, major questions remain about optimizing the risk/benefit profile of LTOT, including: how to best engage patients voluntarily in this process; the safety, tolerability and effectiveness of newer treatment approaches; and optimal treatment selection. The primary objective of the proposed study is to begin to systematically address gaps in this important area to improve pain, reduce risk, and improve quality of life for individuals on LTOT.

ELIGIBILITY:
Inclusion criteria:

Age >/= 18 years

English-speaking

On LTOT, defined as taking daily prescription opioid therapy for 90 days or more

Past week average morphine equivalent dose (MED) >/= 20mg

Willing and able to complete written informed consent

Willing and able to use a mobile/cell phone

Have at least one additional risk for opioid toxicity or overdose from the following list:

Opioid Toxicity or Overdose Risks:

1. Taking benzodiazepines with opioids
2. Substance Use Disorder diagnosis [non-tobacco; Opioid Risk Tool]

2) Having ever experienced an overdose 4) Current major medical problem [e.g. mod-severe liver disease, pancreatitis, chronic pulmonary disease, untreated sleep apnea, hospitalized for an acute medical issue in the past 6 months]a,b 5) Response to BPI Item 8 <30%, suggesting less than moderately clinically meaningful response to pain treatmentc 6) Co-morbid psychiatric diagnosis [Opioid Risk Tool] 7) Signs of opioid misuse [any score >0 on the following COMM Items: 3,4,5,9,10,11,14,15,16] 8)Opioid Risk Tool >3 or Current Opioid Misuse Measure ≥ 9 9) Struggling with any of the following side effects from opioids [self-report]

1. Dizziness and/or falls
2. Difficult-to-manage stomach pain, nausea, constipation or GI issues
3. Fatigue or low energy
4. Sleepiness or sedation
5. Trouble with memory or thinking clearly [COMM Item 1>0]
6. Other troublesome side effect [open answer]

Exclusion criteria:

Known allergy to buprenorphine

Active moderate or severe substance use disorder with the exception of those listed below:

1. . Those with nicotine use disorder.
2. . Those meeting criteria for prescription opioid use disorder using only prescribed opioids will be considered on a case-by-case basis.

Cognitive disorder limiting ability to consent or fully participate in the brief cognitive intervention

Receiving methadone or buprenorphine treatment for OUD or pain

Taking naltrexone

Pregnancy

Currently incarcerated

Taking medications that prolong QTc interval, as determined by study investigators

Personal/immediate family history of Long QT Syndrome.

Significant or unstable condition/s or treatments that may impact safe participation in the study (as determined by the study investigators) such as significant cardiac condition (e.g. poorly-controlled heart failure, current or past cardiac arrhythmia, sustained systolic blood pressure >180), significant metabolic disorder (e.g. labile diabetes, significant electrolyte abnormality), cancer (e.g. brain cancer, chemotherapy-induced cognitive impairment), major psychiatric disorder (e.g. active bipolar disorder, schizophrenia spectrum or other psychotic disorder, suicidal/homicidal intent within the past month, or any suicide attempts within the past year or current active suicidal ideation, as determined by medical clinician), developmental disorder (e.g. autism spectrum disorder, intellectual disability), or other neurologic disease (e.g. movement disorder, multiple sclerosis, moderate to severe brain injury).

Enrolled in a clinical trial or has received an investigational medication or device in the last 30 days.

TMS contraindications (e.g., ferromagnetic implants, conditions or treatments that lower seizure threshold, taking contraindicated medications, no identifiable motor threshold, as determined by study investigators).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Buprenorphine Tolerability | up to Day-13
  Tolerability of open-label transdermal buprenorphine. Buprenorphine tolerability defined as the proportion of patients who do not discontinue buprenorphine due to adverse effects or intolerance.
Pain Severity -with Buprenorphine Patch | up to Day-20
  Pain severity is measured by the Brief Pain Inventory (BPI) Severity Scale and is typically scored as the mean of the four severity items ("average," "worst," "usual," "now," range 0-10) with a higher score being worse.

SECONDARY OUTCOMES:
Buprenorphine Transition Rate | Day-20
  Buprenorphine transition rate defined as the proportion of participants who spontaneously elect to continue buprenorphine after Phase I.
Quality of Life -with Buprenorphine Patch | up to Day-20
  Patient-Reported Outcomes Measurement Information System (PROMIS)-Preference (PROPr) score summarizes multiple domains into a single score anchored at 0 (as bad as dead) and 1 (perfect or ideal health). This score quantifies the value that individuals place on different states of health.
  PROPr is calculated from the scores for the 7 PROMIS domains: Cognition, Depression, Fatigue, Pain Interference, Physical Function, Sleep Disturbance, and Ability to Participate in Social Roles and Activities.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Barth, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States